CLINICAL TRIAL: NCT05566444
Title: Effects of Heat-evoked Experimental Pain on Brain Connectivity
Brief Title: TMS-evoked Potentials During Heat Pain
Acronym: TMS-EEG-heat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Enrico De Martino, Dr, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20220018
Record Dates: First submitted 2022-09-27; First posted 2022-10-04 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Heat; Pain; Electroencephalography; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental heat pain (Experimental): For each participant, we will collect TMS-EEG responses in 4 conditions: 1) Baseline, 2) Heat pain; 3) warm sensation; 4) post-pain.
  Interventions: Device: Heat stimulus

INTERVENTIONS:
Device: Heat stimulus — Contact heat pain stimulus with a termode set at 46 degrees and contact warm stimulus with a termode set at 40 degrees

SUMMARY:
This study investigates the modification of the local-to-global connectivity pattern in response to experimental heat pain. Transcranial magnetic stimulation (TMS) will be applied to elicit electroencephalography (EEG) responses in healthy volunteers. The TMS-evoked potentials (TEPs) will be recorded and serve as a reflection of cortical reactivity to TMS. A thermal cutaneous heat stimulus will induce painful sensations.

DETAILED DESCRIPTION:
Abnormal connectivity patterns interfere with the normal function of a given neuronal network, thus leading to circuit dysfunction and, subsequently, chronic pain. In the last few years, neuroscience has been heavily influenced by network science. This synergistic association provided a new framework for understanding brain function in health and how dysfunction in specific neuronal brain circuits can lead to symptoms. A network comprises nodes (e.g., areas of the brain) and edges (functional connections between nodes). An effective network can process and share large amounts of information while maintaining specificity and not allowing noise to contaminate the flow of information across the circuits. The network approach to brain functioning has been able to integrate what has been known for several decades as spatial structural anatomy with the time-varying streaming of information (connectivity) in a dynamic perspective. In this context, symptoms of diseases are seen as being correlated with specific network abnormalities, and therapeutic interventions as being associated with the normalisation of these abnormal patterns of connection. This study will investigate the responses of specific neuronal brain circuits to experimental heat pain in healthy volunteers. It has been hypothesised that the local-to-global connectivity pattern obtained by the stimulation of different cortical hubs (e.g., the primary motor and dorsolateral prefrontal cortices) will be described by TMS-EEG responses in healthy individuals, and the modification in cortical connectivity in experimental models will be described and compared it with a non-painful sensory stimulation of the same salience.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Speak and understand English

Exclusion Criteria:

* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate
* History of chronic pain or current acute pain
* Contraindications to rTMS application (history of epilepsy, metal in the head or jaw etc.).
* Failure to pass the "TASS questionnaire" (TASS = Transcranial Magnetic Stimulation Adult Safety Screen)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Cortical connectivity | Reduced cortical connectivity (more local) during heat pain. Changes will be investigated before and after heat pain (1 hour)
  Global and local mean field amplitude

SECONDARY OUTCOMES:
Cortical excitability | Reduced cortical excitability during heat pain. Changes will be investigated before and after heat pain (1 hour)
  TMS-evoked potentials

CONTACTS AND LOCATIONS:
Locations (1):
- Enrico De Martino, Aalborg, Denmark